CLINICAL TRIAL: NCT04335396
Title: Screening Patients With Diabetes Mellitus for the Presence of Scleredema Adultorum of Buschke and Characterize Clinical-laboratory Findings of the Newly Identified Cases: a Single-center, Prospective, Obsevational Study
Brief Title: Screening Patients With Diabetes Mellitus for the Presence of Skin Disorder of Scleredema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, dr Varjú Cecília, Associate Professor, MD, PhD, University of Pecs
Other Study IDs: 22400-5/2018 EÜIG
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus; Diabetes Complications; Scleroderma-Like Changes; Scleredema Adultorum
Keywords: Scleredema; Scleroderma-like conditions; Dyslipidemia; NAFLD; Metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Scleredema Adultorum; Dyslipidemias; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with diabetes mellitus: Subgroup 1 - consecutive patients with diabetes mellitus with scleredema skin disorder Subgroup 2 - consecutive patients with diabetes mellitus without scleredema Subgroup 3 - patients with diabetes and scleredema - already cared in the tertiary center of the Rheumatology Department of the University of Pécs, in Hungary.

SUMMARY:
Scleredema is a scleroderma-like skin disorder appearing in 2.5-14% among patients with type 1 or 2 diabetes mellitus. This is a single centre study to screen consecutive patients with diabetes mellitus for the presence of scleredema,and to compare the clinical-laboratory data of patients with and without scleredema. Metabolic and vascular complications of these patients will be focused on.

DETAILED DESCRIPTION:
Scleredema adultorum of Buschke is a scleroderma-like skin disorder characterized by thickened skin with edema in patients' neck, shoulders and back. Graff described three types of scleredema. The first type occurs usually in children after an infection, the second type often associated with haematological malignancies and the third type usually develops in patients with long lasting uncontrolled diabetes mellitus. These patients with diabetes are often obese and have vascular complications. Based on two large cohorts, the prevalence of scleredema among patients with diabetes mellitus was 2.5-14.0% .

The aims of this study is to screen consecutive patients with diabetes mellitus for the presence of scleredema skin disorder and to investigate and compare the clinical-laboratory data of patients with and without scleredema. Both the vascular complications in case history and the parameters of lipid and carbohydrate metabolism will be focused on. All findings will also be compared to another cohort of scleredema-diabetes patients who already treated in our tertiary clinical centre of the University of Pécs in Hungary.

Participants and methods:

About 150 consecutive patients with diabetes mellitus are planned to be investigated. Scleredema skin disorder will be screened by palpation of skin on the nape of the neck, the whole trunk and the shoulders by at least two physicians. Newly recognized patients will be asked to give their consent for undergoing skin biopsy.

Planned clinical examinations and biochemical data collection are as follows:

Besides taking case history, patients will have a complete physical examination, and they will be asked to respond some standardized questions about their diabetes-related earlier vascular and neurological complications, as well as about their skin status.

Repeated blood pressure, measuring weight and their height for defining BMI, for the diagnosis of polyneuropathy neurological physical examination, electroneuronography and calibrated tuning-fork test will be done. Retinopathy will be considered based on ophthalmological examination.

Laboratory investigations are planned including blood count, routine chemistry, glycated haemoglobin (HbA1c), parameters of lipid metabolism as well as thyroid stimulating hormone (TSH) test, unless the patient already had results for these particular lab tests less than three months before. Significant nephropathy will be recorded based on values lower than 60 ml/min/1.73m2 of estimated glomerular filtration rate (eGFR) or the presence of microalbuminuria (>300 mg/die). Calculating of Hepatic steatosis index (HSI) and Framingham steatosis index (FrSI) for define the presence of non-alcoholic fatty liver disease (NAFLD) are also planned.

Statistical analysis of the results will be performed: The distribution of variables planned to be evaluated based on Kolmogorov-Smirnov's test. Comparisons of the values of clinical data between groups will be performed by using a Kruskal-Wallis test for non-parametric data or a one-way ANOVA test for normally distributed continuous variables; Bonferonni's post hoc tests will be used in all cases. Chi-square test or Fisher's test will be used for categorical variables. Clinical-laboratory parameters associated with developing scleredema skin disorder are planned to defined by binary logistic regression with stepwise selection. Statistical analyses will be performed with IBM SPSS Statistics v 24.0 software package (IBM's Corporate, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of diabetes mellitus is based on the criteria of the World Health Organization (WHO), 2006.

The duration of diabetes mellitus must be longer than one year.

Exclusion Criteria:

Patients taking any forms of glucocorticoids in the previous year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
presence of atherogen dyslipidemia | during the whole study, 60 months
  elevated triglycerides (≥1.7 mmol/l) and decreased HDL-cholesterol (<1.03 mmol/l in males and <1.29 mmol/l in females) in the sera
presence of incresed non-HDL cholesterol level of the sera | during the whole study, 60 months
  Serum non-HDL cholesterol was calculated by subtracting HDL-cholesterol from the total cholesterol levels of the sera.

SECONDARY OUTCOMES:
Hepatic steatosis index | during the whole study, 60 months
  8×(alanine aminotransferase/aspartate aminotransferase (ALT/AST) ratio) + BMI (+2, if female; +2, if diabetes mellitus)
Number of vascular complications in patients' medical histories, earlier, than our investigation time | during the whole study, 60 months
  Prevalence of stroke, myocardial infarction, macroangiopathy, nephropathy and retinopathy. neuropathy
Prevalence of polyneuropathy | during the whole study, 60 months
  assessed by electroneuronography

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Varju, MD, PhD, Study Chair — Dept. Rheumatology and Immunology, University of Pécs, Hungary
Locations (1):
- Dept. Rheumatology and Immunology, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sattar MA, Diab S, Sugathan TN, Sivanandasingham P, Fenech FF. Scleroedema diabeticorum: a minor but often unrecognized complication of diabetes mellitus. Diabet Med. 1988 Jul-Aug;5(5):465-8. doi: 10.1111/j.1464-5491.1988.tb01030.x. PMID 2970922
- [Background] Scholz GH, Hanefeld M. Metabolic Vascular Syndrome: New Insights into a Multidimensional Network of Risk Factors and Diseases. Visc Med. 2016 Oct;32(5):319-326. doi: 10.1159/000450866. Epub 2016 Oct 7. PMID 27921043
- [Background] Lee JH, Kim D, Kim HJ, Lee CH, Yang JI, Kim W, Kim YJ, Yoon JH, Cho SH, Sung MW, Lee HS. Hepatic steatosis index: a simple screening tool reflecting nonalcoholic fatty liver disease. Dig Liver Dis. 2010 Jul;42(7):503-8. doi: 10.1016/j.dld.2009.08.002. Epub 2009 Sep 18. PMID 19766548
- [Result] Knobler R, Moinzadeh P, Hunzelmann N, Kreuter A, Cozzio A, Mouthon L, Cutolo M, Rongioletti F, Denton CP, Rudnicka L, Frasin LA, Smith V, Gabrielli A, Aberer E, Bagot M, Bali G, Bouaziz J, Braae Olesen A, Foeldvari I, Frances C, Jalili A, Just U, Kahari V, Karpati S, Kofoed K, Krasowska D, Olszewska M, Orteu C, Panelius J, Parodi A, Petit A, Quaglino P, Ranki A, Sanchez Schmidt JM, Seneschal J, Skrok A, Sticherling M, Sunderkotter C, Taieb A, Tanew A, Wolf P, Worm M, Wutte NJ, Krieg T. European dermatology forum S1-guideline on the diagnosis and treatment of sclerosing diseases of the skin, Part 2: Scleromyxedema, scleredema and nephrogenic systemic fibrosis. J Eur Acad Dermatol Venereol. 2017 Oct;31(10):1581-1594. doi: 10.1111/jdv.14466. Epub 2017 Aug 8. PMID 28786499
- [Result] Cole GW, Headley J, Skowsky R. Scleredema diabeticorum: a common and distinct cutaneous manifestation of diabetes mellitus. Diabetes Care. 1983 Mar-Apr;6(2):189-92. doi: 10.2337/diacare.6.2.189. PMID 6851809
- [Derived] Csonka V, Bodis B, Kovacs D, Farkas N, Kalman E, Czirjak L, Varju C. Screening for the presence of scleroedema adultorum of Buschke in patients with diabetes mellitus: newly diagnosed patients had a high prevalence of dyslipidaemia. Lipids Health Dis. 2021 May 5;20(1):47. doi: 10.1186/s12944-021-01473-1. PMID 33952255